CLINICAL TRIAL: NCT03469934
Title: Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients With Severe Eosinophilic Asthma
Brief Title: Proof of Concept Study to Investigate Etokimab (ANB020) Activity in Adult Participants With Severe Eosinophilic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB020-004; 2017-000647-40 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-04

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etokimab (Experimental): Participants received a single dose of 300 milligrams (mg) etokimab administered on Day 1 by intravenous (IV) infusion over 1 hour. After completing the Day 1 assessments, all participants were followed up for 18 weeks.
  Interventions: Biological: Etokimab
- Placebo (Placebo Comparator): Participants received a single dose of placebo (0.9% sodium chloride) administered on Day 1 by IV infusion over 1 hour. After completing the Day 1 assessments, all participants were followed up for 18 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Etokimab — Administered on Day 1 over 1 hour by IV infusion
  Other Names: ANB020
  Arms: Etokimab
Drug: Placebo — Administered on Day 1 over 1 hour by IV infusion
  Arms: Placebo

SUMMARY:
This is a proof of concept study designed to assess the effects of a single intravenous dose of etokimab compared to placebo in adult participants with severe eosinophilic asthma. This study will also assess the safety and tolerability of etokimab in adult participants with severe eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed clinical diagnosis of eosinophilic asthma
* History of diagnosis of eosinophilic asthma
* Severe asthma diagnosed according to the Global Initiative for Asthma (GINA) 2016
* Body mass index (BMI) of 18 to 38 kilograms per squared meters (kg/m^2) (inclusive) and total body weight > 50 kg (110 pounds)
* Women of childbearing potential must have a negative serum pregnancy test at screening and be willing to use highly effective methods of contraception throughout the study
* Male participants must be willing to use effective methods of contraception during the entire study period.
* Participant must be on high dose inhaled corticosteroids (ICS) plus long-acting beta-2-agonists (LABA)
* Willing and able to comply with the study protocol requirements
* Have the ability to read and understand the study procedures and can communicate meaningfully with the Investigator and staff

Exclusion Criteria:

* Have concomitant medical condition(s) which may interfere with the Investigator's ability to evaluate the participant's response to the investigational product (IP)
* Have experienced severe life threatening anaphylactic reactions
* Have received any IP within a period of 3 months or 5 half lives of an IP
* Have received high dose systemic corticosteroids
* Have received treatment with biologics, such as mepolizumab or omalizumab, within 3 months or 5 half lives (whichever is longer) before screening
* Abnormal electrocardiogram (ECG) assessment at screening
* Uncontrolled hypertension, or acute ischemic cardiovascular diseases
* If female, is pregnant or lactating, or intend to become pregnant during the study period
* History (or suspected history) of alcohol or substance abuse within 2 years before screening
* Any comorbidity that the Investigator believes is a contraindication to study participation
* Have any other physical, mental, or medical conditions which, in the opinion of the Investigator, make study participation inadvisable or could confound study assessments
* Planned surgery during the study or 30 days before screening
* History of malignancy within 5 years, except non melanoma skin cancer which has been fully treated with no current active disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Randazzo, MD, Study Director — AnaptysBio, Inc.
Locations (7):
- United States (4):
  - Midwest Allergy Sinus Asthma, Normal, Illinois
  - Pulmonary & Critical Care Specialists, Novi, Michigan
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Allergy & Asthma Center of Southern Oregon, Medford, Oregon
- United Kingdom (3):
  - Medicines Evaluation Unit, Manchester, Greater Manchester
  - Glenfield Hospital, Leicester, Leicestershire
  - Churchill Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pavord ID, Marquette A, Kahm P, Pinkstaff J, Sacco N, Londei M. Single-dose Phase 2a trial of etokimab (anti-IL-33) in severe eosinophilic asthma. Paper presented at the European Academy of Allergy and Clinical Immunology (EEACI) Congress 2019; June 1-5, 2019; Lisbon, Portugal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 centers in the United Kingdom (UK) and United States of America (USA).
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to receive a single dose of either etokimab or placebo.
Period: Overall Study
Arm/Group | Etokimab | Placebo
Started | 12 | 13
Pharmacodynamic (PD) Analysis Set (All participants who received etokimab or placebo and provided at least one evaluable post-dose PD measurement without any events or protocol deviation deemed to affect PD assessment.) | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received etokimab or placebo.
Groups:
- Etokimab: Participants received a single dose of 300 mg etokimab administered on Day 1 by IV infusion over 1 hour. After completing the Day 1 assessments, all participants were followed up for 18 weeks.
- Total: Total of all reporting groups
Arm/Group | Etokimab | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.72) | 36.3 (14.70) | 38.4 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eosinophil Count [Mean (Standard Deviation); unit: 10^9 cells/Liters] | 0.545 (0.379) | 0.705 (0.362) | 0.628 (0.3715)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peripheral Eosinophil Count at Day 22
Time Frame: Baseline, Day 22
Population: Participants in the PD analysis set with available data were evaluated.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/Liters
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 11 | 13
10^9 cells/Liters | -0.199 [-0.351 to -0.046] | -0.141 [-0.280 to -0.002]
Statistical Analysis 1: Comparison: Etokimab vs Placebo; Mixed-model repeated measures (MMRM) analysis with fixed terms for treatment, time point of measurement, and treatment by time point interaction, baseline eosinophil count as a covariate, and a repeated time point effect within a participant; Test type: Other; p = 0.5703, Mixed-model repeated measures; Least Squares (LS) Mean Difference = -0.058, 95% CI 2-sided [-0.265 to 0.150]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
  An AE was considered "serious" if there was any of the following outcomes: death, life-threatening, Inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of ability to conduct normal life functions, congenital anomaly/birth defect, other important medical events.
  Treatment-emergent adverse events (TEAEs) were defined as AEs that started or worsened in severity on or after the date and time of the study drug infusion.
Time Frame: From first dose to Day 127
Population: Participants in the safety analysis set were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 13
Participants
  Any TEAEs | 6 | 5
  Serious TEAEs | 0 | 0

3. Primary Outcome: Number of Asthma Exacerbations
Description: Asthma exacerbation was defined as follows:
  1. Use of systemic corticosteroids (or a temporary increase in a stable oral corticosteroid background dose) for at least 3 days; a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of systemic corticosteroids.
     OR
  2. An emergency room/urgent care visit (defined as evaluation and treatment for <24 hours in an emergency department or urgent care center) due to asthma that required systemic corticosteroids (as per above).
     OR
  3. An inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours due to asthma).
Time Frame: From first dose to Day 127
Population: Full analysis set included all participants who received etokimab or placebo and had at least one post-baseline blood eosinophils count assessment.
Measure: Number; unit: asthma exacerbations
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 13
asthma exacerbations | 1 | 1

4. Primary Outcome: Number of Participants With Positive Anti-drug Antibody
Time Frame: Day 1, Day 8, Day 36, Day 85, Day 106, end of study (up to Day 127)
Population: Participants in the safety analysis set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Day 1 | 1 | 1
  Day 8 | 0 | 2
  Day 36 | 0 | 2
  Day 85 | 1 | 1
  Day 106 | 1 | 1
  End of Study (up to Day 127) | 2 | 1

5. Secondary Outcome: Change From Baseline in Peripheral Eosinophil Count at Day 127
Time Frame: Baseline, Day 127
Population: Participants in the PD analysis set were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/Liters
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 13
10^9 cells/Liters | -0.194 [-0.330 to -0.058] | -0.144 [-0.275 to -0.014]
Statistical Analysis 1: Comparison: Etokimab vs Placebo; MMRM analysis with fixed terms for treatment, time point of measurement, and treatment by time point interaction, baseline eosinophil count as a covariate, and a repeated time point effect within a participant; Test type: Other; p = 0.5901, Mixed-model repeated measures; LS Mean Difference = -0.050, 95% CI 2-sided [-0.239 to 0.139]

6. Secondary Outcome: Change From Baseline in Prebronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Day 127
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Baseline, Day 127
Population: Participants in the full analysis set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 12
Liters | 0.27 [0.03 to 0.51] | 0.18 [-0.06 to 0.42]
Statistical Analysis 1: Comparison: Etokimab vs Placebo; Change from baseline for FEV1 was compared between etokimab and placebo using an analysis of covariance (ANCOVA) with treatment as fixed effect and baseline result as covariate and participant as a random effect; Test type: Other; p = 0.5960, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-0.25 to 0.43], Standard Error of Mean 0.164

7. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) at Day 127
Description: Measurement of FeNO was performed in accordance with the guidelines published by American Thoracic Society/European Respiratory Society (ATS/ERS).
Time Frame: Baseline, Day 127
Population: Participants in the full analysis set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: parts per billion
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 12 | 12
parts per billion | 2.10 [-11.59 to 15.78] | -0.43 [-14.12 to 13.25]
Statistical Analysis 1: Comparison: Etokimab vs Placebo; Change from baseline for FeNO was compared between etokimab and placebo using an ANCOVA with treatment as fixed effect and baseline result as covariate and participant as a random effect; Test type: Other; p = 0.7993, ANCOVA; LS Mean Difference = 2.53, 95% CI 2-sided [-17.90 to 22.96], Standard Error of Mean 9.823

8. Secondary Outcome: Change From Baseline in Whole Blood Ex-vivo Induced Interferon Gamma (IFN-γ)
Description: Blood samples for ex vivo induced IFN-γ assessment were collected in a sodium heparin tube. The measurement of ex vivo induced IFN-γ was performed using validated assay method.
Time Frame: Baseline, Day 8, Day 36, Day 85, Day 106, and End of Study (up to Day 127)
Population: Participants in the PD analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | Etokimab | Placebo
Number analyzed (Participants) | 4 | 4
nanograms per liter (ng/L)
  Baseline | 702.215 (581.947) | 2490.575 (3577.893)
  Change at Day 8: number analyzed (Participants) | 3 | 2
  Change at Day 8 | -377.747 (359.751) | NA (NA) — The mean and standard deviation were not determined as the values were below the lower limit of quantification (LLOQ).
  Change at Day 36: number analyzed (Participants) | 2 | 3
  Change at Day 36 | NA (NA) — The mean and standard deviation were not determined as the values were below the lower limit of quantification (LLOQ). | 5035.623 (5790.397)
  Change at Day 85: number analyzed (Participants) | 2 | 1
  Change at Day 85 | NA (NA) — The mean and standard deviation were not determined as the values were below the lower limit of quantification (LLOQ). | NA (NA) — The mean and standard deviation were not determined as the values were below the lower limit of quantification (LLOQ).
  Change at Day 106: number analyzed (Participants) | 2 | 0
  Change at Day 106 | NA (NA) — The mean and standard deviation were not determined as the values were below the lower limit of quantification (LLOQ). |
  Change at end of study (up to Day 127) | 401.108 (1002.500) | 2635.555 (4491.890)

9. Secondary Outcome: Maximum Observed Concentration (Cmax) of Etokimab
Description: Cmax was obtained directly from the observed concentration versus time data.
Time Frame: pre-dose, 0.50 hours post-start of infusion, end of infusion (EOI), EOI+3 hours, EOI+6 hours, and then 24, 168, 504, 840, 1512 hours post-start of infusion
Population: Pharmacokinetic (PK) analysis set included all participants who received etokimab and have at least one post-dose serum concentration data value available for etokimab without any events or protocol deviation deemed to affect PK assessments.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Etokimab
Number analyzed (Participants) | 11
micrograms per milliliter (µg/mL) | 79.84 (20.52)

10. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Etokimab
Description: Tmax was obtained directly from the observed concentration versus time data.
Time Frame: pre-dose, 0.50 hours post-start of infusion, EOI, EOI+3 hours, EOI+6 hours, and then 24, 168, 504, 840, 1512 hours post-start of infusion
Population: Participants in the PK analysis set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Etokimab
Number analyzed (Participants) | 11
hours | 1.020 [0.53 to 4.08]

11. Secondary Outcome: Area Under the Concentration-time Curve in Serum From Time Zero (Predose) Extrapolated to Infinite Time (AUC0-inf) of Etokimab
Description: AUC0-inf was calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the apparent terminal rate constant.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: hours*µg/mL
Arm/Group | Etokimab
Number analyzed (Participants) | 11
hours*µg/mL | 14400 (4698)

12. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of Etokimab
Description: AUC0-last was calculated by linear up/log down trapezoidal summation.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: hours*µg/mL
Arm/Group | Etokimab
Number analyzed (Participants) | 11
hours*µg/mL | 13590 (4117)

13. Secondary Outcome: Apparent Total Body Clearance (CL) of Etokimab
Description: CL was calculated as dose/ AUC0-inf.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Etokimab
Number analyzed (Participants) | 11
L/hour | 0.02278 (0.006896)

14. Secondary Outcome: Apparent Terminal Rate Constant (λz) of Etokimab
Description: λz was determined by linear regression of the terminal points of the log-linear concentration-time curve.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Etokimab
Number analyzed (Participants) | 11
1/hour | 0.002174 (0.0006052)

15. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Etokimab
Description: Apparent terminal half-life was determined as (natural logarithm of 2 [ln2] divided by λz).
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Etokimab
Number analyzed (Participants) | 11
hours | 343.3 (102.5)

16. Secondary Outcome: Volume of Distribution During Terminal Phase (Vz) of Etokimab
Description: Vz was estimated by dividing the systemic clearance by λz.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Etokimab
Number analyzed (Participants) | 11
Liters | 10.55 (1.701)

17. Secondary Outcome: Volume of Distribution at Steady State Following Intravenous Dosing (Vss) of Etokimab
Description: Volume of distribution at steady state following intravenous dosing was calculated as [([AUMClast + ([tlast*Clast]/λz) + Clast/λz^2]/ AUC(0-inf)) - TI/ 2]*CL, Clast is last observed (quantifiable) plasma concentration, where AUMClast is the area under the moment curve from the time of dosing to Clast, tlast is the time of Clast, and TI is infusion duration.
Time Frame: as for outcome 10
Population: Participants in the PK analysis set were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Etokimab
Number analyzed (Participants) | 11
Liters | 8.485 (1.378)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 127
Description: Participants from the Safety Analysis Set were analyzed.
Arm/Group | Etokimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 6/12 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etokimab (N=12) | Placebo (N=13)
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03469934/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03469934/SAP_001.pdf